CLINICAL TRIAL: NCT02088996
Title: Electrical Stimulation and Chemotherapy Induced Peripheral Neuropathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Studie 3
Record Dates: First submitted 2014-03-10; First posted 2014-03-17 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IT and LWD on high power (Active Comparator): IT and LWD on high power
  Interventions: Device: longwave diathermy on high power and interferential therapy
- LWD on low power (Placebo Comparator): LWD on low power
  Interventions: Device: longwave diathermy on low power

INTERVENTIONS:
Device: longwave diathermy on high power and interferential therapy
  Arms: IT and LWD on high power
Device: longwave diathermy on low power
  Arms: LWD on low power

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) implies sensory or deficits pain, loss of motor functions and impaired proprioception which in turn may affect balance and fine motor skills. It is mainly subjected to the peripheral parts of the extremities, may be transient or permanent.CIPN is a common, potentially severe and often dose-limiting side effect after patient exposure of numerous classes of antineoplastic agents including platins, taxanes, vinca alkaloids, bortezomib and thalidomide. At present, no evidence based treatment of CIPN is available. A variety of different drugs or drug combinations have been clinically tested but the value of these treatments is uncertain. Many patients with CIPN are referred to physiotherapy but still this treatment is more based on clinical experience and tradition than scientific evidence. In a nonrandomized study, sensory electrical stimulation(MC5-A Calmare ®) was tested on 16 persons.The electrodes were placed on the hand and foot and intensity was gradually increased and given daily for 10 days. Pain was reduced 20% in numeric pain score for 15 of the 16 participating patients.

Our clinical experience indicates that treatment with long wave diathermy (LWD) may decrease CIPN symptoms. This treatment produces electromagnetic radiation according the capacitor method with heightened circulation and heat which is assumed to reduce pain. Interferential Therapy (IT) is an electro-physical method which is based on an electric field in the painful area through four electrodes or vacuum cups placed on the skin. Increased blood circulation and pain relief is supposed to be achieved. IT use two different intermediate frequencies (1001-10000 Hz) alternating currents in the painful area. The treatment effect correspond to the "gate control-theory"; inhibition of pain signals in small diameter fibers by activity in large-diameter Aβ-fibers by spinal neurons. Some studies have shown effect in treating pain with interferential currents when pain is experimentally induced or induced by cold in otherwise pain-free volunteers, when compared to a control or placebo.

The hypothesis of this study is that the combination therapy longwave diathermy on high power and interferential currents gives better results than longwave diathermy on low power.

DETAILED DESCRIPTION:
A randomized controlled trial to investigate the effects of combination therapy longwave diathermy on high power and interferential currents, as compared to longwave diathermy at low power (control group) for sensory and motor symptoms in patients with CIPN in the feet and lower legs. Sensory and motor symptoms are defined as numbness, pain, discomfort and balance impairment.

Interferential currents is administered by "Electrostimulation unit ES-520 & Vacuum Unit.

The longwave diathermy at low and high power is given thru capacitive energy transfer system and is administered by "Skanlab 25 Bodywave".

The drugs that have been clinically tested in other studies were magnesium, calcium, vitamin E and B6, glutamine, glutathione, n-acetyl cysteine omega-3 fatty acids, acetyl-L-carnitine and alpha lipoic acid.

ELIGIBILITY:
Inclusion Criteria:

- patients over 18 years who received chemotherapy and had documented side effects such as numbness, tingling, pain or swelling sensation in the feet/lower legs.

Exclusion Criteria:

* pregnancy, thrombosis thrombophlebitis in the feet or lower legs, muscle cramps, acute bleeding disorders, dementia, type 1 diabetes mellitus, open sores on the feet or lower legs, peripheral sensory neuropathies due to causes other than chemotherapy, ongoing chemotherapy with drugs known to cause CIPN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in numbness from baseline | baseline and 12 weeks
  The definition of spreading of numbness was pins and needles, tingling and parasthesias. Patients were asked to draw the distribution of their numbness in their legs and feet on a sketch, -which was constructed based on pain drawing sketch.

SECONDARY OUTCOMES:
Change in pain intensity and discomfort from baseline . | baseline and 12 weeks
  Numerical rating scale (NRS) were used for measuring the intensity of pain. This is a reliable instrument and has been validated for patients with cancer. Patients rate their pain from zero to 100, with zero reflecting no pain and 100 reflecting the worst possible pain. Discomfort is defined as uncomfortable not knowing where your feet are in relation to the room and met with NRS.
Change in numbness from baseline | baseline and 6 months
  The definition of spreading of numbness was pins and needles, tingling and parasthesias. Patients were asked to draw the distribution of their numbness in their legs and feet on a sketch, -which was constructed based on pain drawing sketch.
Change in pain intensity and discomfort from baseline | baseline and 6 months
  Numerical rating scale (NRS) were used for measuring the intensity of pain. This is a reliable instrument and has been validated for patients with cancer. Patients rate their pain from zero to 100, with zero reflecting no pain and 100 reflecting the worst possible pain. Discomfort is defined as uncomfortable not knowing where your feet are in relation to the room and met with NRS.

OTHER OUTCOMES:
Change in balance ability/disability from baseline | baseline and 12 weeks
  1. Romberg test (standing with both ankle bones touching each other with the hands crossed and touching the shoulders, max time 30 seconds) as well as, tightened Romberg test (tandem standing with with the hands crossed and touching the shoulders, max 60 seconds).
  2. One-legged stance test (standing on one leg with the hands crossed and touching the shoulders, max 30 seconds). These tests have good validity and reliability when tested on healthy elderly females.
  The patient had three attempts of each test of which the best attempt was recorded. All tests were performed with open and closed eyes. The time was stopped when the patient moved the feet/arms position and/or looked when the eyes should be closed.
Change in quality of life from baseline | baseline and 12 weeks
  Generic health-related quality of life was measured by the European quality of life questionnaire (EQ-5D). The following 5 dimensions are measured: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problem, some problems, extreme problems. (EuroQol-Group, 1990). EQ-5D has shown good reliability and validity when tested in older people (Haywood, Garratt, Fitzpatrick, 2005).
Change in expectations from baseline | baseline and 12 weeks
  Expectations of treatment outcome were evaluated before treatment started on a numerical scale (0-100). The question asked to the patients was: What is your expectation of treatment effect with electroconvulsive therapy at CIPN for spreading of numbness, pain, discomfort, subjective experienced balance and balance? Background data such as age, sex, diagnosis, chemotherapy variety, when chemotherapy started and completed were recorded before treatment.
Change in balance ability/disability from baseline | baseline and 12 weeks
  1. Measurement of subjective experience of balance Dizziness Handicap Inventory was used for measurement of patients experience ot their balance. The questionnaire contains 25 questions and has good reliability in vestibular disorders/disabilities. In this study , however the form was abbreviated and contained only 15 questions, ten questions were omitted since they were considered to be inappropriate for this patient group.
  2. Activities-Specific Balance Confidence Scale (ABC) is a subjective measure of confidence in performing various ambulatory activities without falling. It is a 16-item self-report measure in which patients rate their balance confidence in performing several activities. Each item is rated on a 0-100 scale. Zero represents no confidence; a score of 100 represents complete confidence. The instrument is validated and demonstrated good test-retest reliability on elderly persons.
Change in quality of life from baseline | baseline and 6 months
  Generic health-related quality of life was measured by the European quality of life questionnaire (EQ-5D). The following 5 dimensions are measured: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problem, some problems, extreme problems. (EuroQol-Group, 1990). EQ-5D has shown good reliability and validity when tested in older people (Haywood, Garratt, Fitzpatrick, 2005).
Change in expectations from baseline | baseline and 6 months
  Expectations of treatment outcome were evaluated before treatment started on a numerical scale (0-100). The question asked to the patients was: What is your expectation of treatment effect with electroconvulsive therapy at CIPN for spreading of numbness, pain, discomfort, subjective experienced balance and balance? Background data such as age, sex, diagnosis, chemotherapy variety, when chemotherapy started and completed were recorded before treatment.
Change in balance ability/disability from baseline | baseline and 6 months
  1. Measurement of subjective experience of balance Dizziness Handicap Inventory was used for measurement of patients experience ot their balance. The questionnaire contains 25 questions and has good reliability in vestibular disorders/disabilities. In this study , however the form was abbreviated and contained only 15 questions, ten questions were omitted since they were considered to be inappropriate for this patient group.
  2. Activities-Specific Balance Confidence Scale (ABC) is a subjective measure of confidence in performing various ambulatory activities without falling. It is a 16-item self-report measure in which patients rate their balance confidence in performing several activities. Each item is rated on a 0-100 scale. Zero represents no confidence; a score of 100 represents complete confidence. The instrument is validated and demonstrated good test-retest reliability on elderly persons.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Andreasson, MD, Principal Investigator — Västmanlands sjukhus, Västerås
Locations (1):
- Västmanlands sjukhus, Västerås, Onkologiska kliniken, Västerås, Sweden